CLINICAL TRIAL: NCT03533231
Title: Efficiency of Triple Antibiotic Mixture and Propolis as Intracanal Medication in Revascularization Process in Immature Apex: A Clinical Study
Brief Title: Efficiency of Triple Antibiotic Paste, Ciprofloxacin/Propolis, Ciprofloxacin/Metronidazole, Propolis/Metronidazole Combinations on Revascularization Process of Immature Necrotic Maxillary Incisors of Patients 8-18 Years Old.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tariq Yehia (Other)
Responsible Party: Sponsor-Investigator, Tariq Yehia, Lecturer of Endodontics, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECID011508
Record Dates: First submitted 2018-04-24; First posted 2018-05-23 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Dental Pulp Necrosis; Periapical Abscess; Root Canal Infection
Keywords: Pulp regeneration, intracanal medication
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Abscess | interventions — Ciprofloxacin; Propolis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Triple Antibiotic Paste (TAP) (Active Comparator): It consisted of Ciprofloxacin (Ciprocin 250 mg tablets; EPICO, Cairo, Egypt), Metronidazole (Flagyl 500 mg tablets; Sanofi Aventis Pharma, Cairo, Egypt), Doxycycline (Vibramycin 100 mg capsules; Pfizer, Cairo, Egypt). One Doxycycline capsule content was evacuated in a sterile mortar, one tablet of metronidazole and one tablet of ciprofloxacin were crushed and ground in the same mortar using a pestle into homogenous powder. Saline drops (Otrivin baby saline; Novartis, Cairo, Egypt) were added and mixed using the pestle until a creamy paste was achieved (Sabrah et al. 2013, Nagy et al. 2014). TAP was then used for canal disinfection.
  Interventions: Combination Product: Canal Disinfection Triple Antibiotic Paste (TAP)
- Ciprofloxacin + Propolis Paste (Experimental): Ethanol extract of raw propolis (EEP; ElEzaby Co. Labs, Cairo, Egypt.) was prepared by adding 10 gm of propolis (Imtinan, Cairo, Egypt) to 40 gm of 70% ethanol (ElGomhorya Co., Cairo, Egypt) (for 20% tincture) in a dark container to prevent reduction of propolis. The container was sealed and placed at room temperature for a period of three weeks. The sealed container was manually shaken every 2 days to ensure proper mixing. After 3 weeks, the container was opened and ethanol extract of propolis was obtained. Ethanol-free EEP was made by evaporating the ethanol in a water bath. EEP was then mixed with Ciprofloxacin powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved. This paste was then used for canal disinfection.
  Interventions: Combination Product: Ciprofloxacin + Propolis Paste
- Ciprofloxacin + Metronidazole Paste (Active Comparator): Ciprofloxacin powder was mixed with Metronidazole powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved. This paste was then used for canal disinfection.
  Interventions: Combination Product: Ciprofloxacin + Metronidazole Paste
- Propolis + Metronidazole paste (Experimental): Ethanol Extract of Propolis (EEP) was mixed with Metronidazole powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved. This paste was then used for canal disinfection.
  Interventions: Combination Product: Propolis + Metronidazole paste

INTERVENTIONS:
Combination Product: Canal Disinfection Triple Antibiotic Paste (TAP) — Patients were treated as follows: Caries was excavated; access cavity was prepared. The rubber dam was then applied and working length was determined. Canal space was irrigated using 40 cc of NaOCl 2.6% solution and final flush of saline. Canal space was dried using paper points. One cc of the prepared paste was injected into the canals using a sterile plastic syringe with 20" gauge needle. The access cavity was then sealed using temporary restoration. After the 3 weeks, anesthesia without vasoconstrictor was administrated. The antibiotic paste was removed and the canal was irrigated using a sterile saline and dried using paper points. Sterile hand file size #25 was introduced into the root canal beyond the working length to induce bleeding. The bleeding was allowed to reach a 3-mm level below the cemento-enamel junction. MTA was used to seal the root canal at the cervical level. After one week, adhesive composite resin was used to seal the access cavity.
  Arms: Triple Antibiotic Paste (TAP)
Combination Product: Ciprofloxacin + Propolis Paste
  Arms: Ciprofloxacin + Propolis Paste
Combination Product: Ciprofloxacin + Metronidazole Paste
  Arms: Ciprofloxacin + Metronidazole Paste
Combination Product: Propolis + Metronidazole paste
  Arms: Propolis + Metronidazole paste

SUMMARY:
This Study Was Made to Evaluate the Antibacterial Effect of Different Antibacterial Combinations on Revascularization Process in Permanent Anterior Immature Teeth. Immature Necrotic Permanent Maxillary Incisors (n = 40) of Patients 8-18 Years Old Were Divided Into 4 Equal Groups (Each n = 10) According to the Intracanal Medicament: Group 1 Was Treated With Triple Antibiotic Paste (TAP), Group 2 Was Treated With Ciprofloxacin + Propolis Paste (CP), Group 3 Was Treated With Ciprofloxacin + Metronidazole Paste (CM), Group 4 Was Treated With Propolis + Metronidazole Paste (PM). Cases Were Followed at Regular Intervals up to 18 Months Clinically and Radiographically.

DETAILED DESCRIPTION:
Introduction In the last 10 years, numerous published cases and case series described the revascularization or regenerative endodontics. Revascularization is a conservative method for inducing maturogenesis in necrotic immature teeth. The favorable outcomes of regenerative endodontics are largely dependent on the adequate disinfection of the root canal. These canals with compromised fragile underdeveloped dentinal walls represent a contraindication for mechanical instrumentation; thus, chemical debridement remains the main form of disinfection. A mixture of ciprofloxacin, metronidazole, and minocycline, known as the triple antibiotic paste (TAP), has been shown to be very effective in eliminating endodontic pathogens in vitro and in situ. However, TAP has an adverse effect on stem cell survival. Discoloration of the tooth is a problem mostly related to the use of minocycline in TAP. Moreover, TAP can demineralize dentin resulting in reduced microhardness and fracture resistance. Propolis, a flavonoid-rich resinous product of honeybees, is ten times less cytotoxic than calcium hydroxide and has a well-known antibacterial effect. Therefore, creating alternatives to the TAP for disinfecting the root canal of necrotic teeth during the process of pulp revascularization is thought to be of value.

Materials and methods Forty patients with immature, nonvital maxillary incisors were included in this study from the outpatient clinic of the Faculty of Dentistry, Ain Shams University, Cairo, Egypt. A detailed medical and dental history was obtained from each patient's parents or guardians. Only medically free patients were included in this research. The clinical and radiographic exclusion criteria were teeth with vertical fractures, periodontally involved teeth, and nonrestorable teeth. All procedures were performed after obtaining proper institutional review board approval based on the regulations of the Ethical Committee of the Faculty of Dentistry, Ain Shams University. Intraoral periapical radiographs revealed immature apices. The age of the patients ranged between 8 and 18 years. Informed consent was signed for each case by the patient's parents or guardians including the proposed treatment and possible outcomes or complications.

Cases were divided randomly and equally into 4 groups according to the intracanal medicament (10 patients for each group):

TAP group: was treated with Triple Antibiotic Paste CP group: was treated with Ciprofloxacin + Propolis paste CM group: was treated with Ciprofloxacin + Metronidazole paste PM group: was treated with Propolis + Metronidazole paste

1. Triple Antibiotic Paste (TAP):

   It consisted of Ciprofloxacin (Ciprocin 250 mg tablets; EPICO, Cairo, Egypt), Metronidazole (Flagyl 500 mg tablets; Sanofi Aventis Pharma, Cairo, Egypt), Doxycycline (Vibramycin 100 mg capsules; Pfizer, Cairo, Egypt). One Doxycycline capsule content was evacuated in a sterile mortar, one tablet of metronidazole and one tablet of ciprofloxacin were crushed and ground in the same mortar using a pestle into homogenous powder. Saline drops (Otrivin baby saline; Novartis, Cairo, Egypt) were added and mixed using the pestle until a creamy paste was achieved.
2. Ciprofloxacin + Propolis Paste:

   Ethanol extract of raw propolis (EEP; ElEzaby Co. Labs, Cairo, Egypt.) was prepared by adding 10 gm of propolis (Imtinan, Cairo, Egypt) to 40 gm of 70% ethanol (ElGomhorya Co., Cairo, Egypt) (for 20% tincture) in a dark container to prevent reduction of propolis. The container was sealed and placed at room temperature for a period of three weeks. The sealed container was manually shaken every 2 days to ensure proper mixing. After 3 weeks, the container was opened and ethanol extract of propolis was obtained. Ethanol-free EEP was made by evaporating the ethanol in a water bath. EEP was then mixed with Ciprofloxacin powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved.
3. Ciprofloxacin + Metronidazole Paste:

Ciprofloxacin powder was mixed with Metronidazole powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved.

4) Propolis + Metronidazole paste: EEP was mixed with Metronidazole powder in the ratio 1:1. Saline drops were added and mixed using the pestle until a creamy paste was achieved.

A preoperative radiograph was taken using the standardized paralleling technique by the Rinn XCP (Rinn Corporation Elgin, Illinois, USA) alignment system and Fona ScaNeo intra-oral digital imaging system (FONA Dental, Bratislava, Slovak Republic). Patients were treated as follows: Caries was excavated; access cavity was prepared. The rubber dam was then applied and working length was determined with a periapical radiograph taken with a file inserted into the canal. Canal space was debrided using K file size #80. Canal space was irrigated using 40 cc of NaOCl 2.6% solution and final flush of saline. Canal space was dried using paper points. The antibiotic paste was prepared as previously described. One cc of the prepared paste was injected into the canals using a sterile plastic syringe with 20" gauge needle. Care was taken to avoid apical extrusion and to minimize placement in the coronal portion of the tooth. The access cavity was then sealed using temporary restoration (Coltosol F; Coltene Whaledent, Altstatten, Switzerland) over plain cotton. After the 3 weeks, under the same aseptic conditions, anesthesia without vasoconstrictor (Mepecaine, Alexandria Co., Alexandria, Egypt) was administrated. The tooth was re-entered, the antibiotic paste was removed and the canal was irrigated using a sterile saline and dried using paper points.

Sterile hand file size #25 was introduced into the root canal and placed at 2 mm beyond the working length to induce bleeding into the canal. The bleeding was allowed to reach a 3-mm level below the cemento-enamel junction, and teeth were left at rest for 5 minutes so that a blood clot could be formed. Next, a 3-mm plug of MTA (Angelus; Londrina, Brazil) was inserted into the canals using a suitable-sized amalgam carrier to seal the root canal at the cervical level. The MTA plug was verified radiographically. The MTA plug was then covered by moist cotton and temporary filling. After one week, MTA setting was confirmed clinically, adhesive composite resin (Z250 Restorative; 3M ESPE, St Paul, Minnesota, USA) was used to seal the access cavity.

Evaluation:

Patients were recalled for follow up at 3, 6, 9, 12, and 18 months. Follow-up included the clinical assessment of pain and/or swelling and standardized radiographic assessment, which included the following:

1. An increase in root length
2. An increase in root thickness
3. A decrease in apical diameter
4. A change in periapical bone density All radiographic measures were collected by the same investigator. All radiographic measurements were repeated after 1 week, and the mean of the 2 sets was considered as the final value.

Increase in root length: A measuring scale was set in the Image-J software (Image-J v1.44, US National Institutes of Health, Bethesda, MD) by measuring a known clinical dimension to its radiographic dimension. The scale was calculated as number of measured pixels per mm length. Root length was measured as a straight line from the cemento- enamel junction to the radiographic apex of the tooth in millimeters. Pre and follow-up root lengths were measured using Image-J analysis software. Difference in length was calculated. Percentage of increase in length was calculated as follows: percentage of increase in length = [(postoperative length - preoperative length) / preoperative length] X 100.

Increase in root thickness: Using the preset measurement scale, the level of the apical third was determined and fixed from the cemento-enamel junction. The root thickness and the pulp width were measured mesiodistally at this level in millimeters. Mesiodistal dentin thickness was measured by subtraction of the pulp space from the whole root thickness. Pre and follow-up root thicknesses were measured. Measurements were done pre and post operatively at the same fixed level. Difference in dentin thickness was calculated. Percentage of increase in dentin thickness was calculated as follows: percentage of increase in dentin thickness = [(postoperative thickness - preoperative thickness) / preoperative thickness] X 100.

Decrease in apical diameter: Using the preset measurement scale, the mesiodistal diameter of the apical foramen was measured in millimeters. Measurements were done pre and postoperatively. Percentage of apical closure was calculated as follows: percentage of apical closure = [(preoperative apical diameter - postoperative apical diameter) / preoperative apical diameter] X 100.

Periapical bone density:

Periapical bone density was estimated using Image-J software as follows: periapical area was located and analyzed for bone density. Average area density was measured in scale from 0 (black) to 255 (white) and recorded for each radiograph. The same area was then measured in subsequent radiographs and average densities were recorded for the follow up radiographs. The difference between densities was calculated between subsequent radiographs. Percentage of change in density was calculated from the original pre-operative radiograph density as follows: percentage of change in density = [(postoperative bone density - preoperative bone density)/preoperative bone density] X 100.

Data were collected, tabulated and statistically analyzed using statistical analysis software SPSS (Statistical Packages for the Social Sciences 19.0, IBM, Armonk, NY). Two-way analysis of variance was performed. The Tukey post hoc test was used in case of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent anterior teeth having immature apex.
2. Established radiographic periapical pathosis.
3. History of previous trauma.
4. Compliant patient/parent.

Exclusion Criteria:

1. teeth with vertical fractures, periodontally involved teeth, and nonrestorable teeth.
2. Patients with vital teeth.
3. Patients with heart disease or systemic disorders.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in periapical pathosis | baseline, 3 months, 6 months, 9 months, 12 months, and 18 months
  Change in periapical bone density on follow up radiographs
Change in root length | baseline, 3 months, 6 months, 9 months, 12 months, and 18 months
  Change in root length on follow up radiographs
Change in root thickness | baseline, 3 months, 6 months, 9 months, 12 months, and 18 months
  Change in root thickness on follow up radiographs
Change in apical diameter | baseline, 3 months, 6 months, 9 months, 12 months, and 18 months
  Change in apical diameter on follow up radiographs